CLINICAL TRIAL: NCT06253338
Title: Optimization of Radiation Protection Through Genomic Analyses in the Analysis of Changes in Cells of the Hematopoietic System Before and During High Dose External Beam Radiotherapy
Brief Title: Optimization of Radiation Protection Through Genomic Analyses
Acronym: ORtogether
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Essen (Other)
Responsible Party: Principal Investigator, Maja Guberina, PD Dr. med. (MD) / specialist forradiation oncology, senior consultant, University Hospital, Essen
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: 23-11672-BO
Record Dates: First submitted 2023-12-30; First posted 2024-02-12 (Actual); Last update posted 2024-09-27 (Actual); Status verified 2024-09

CONDITIONS: DNA; Cancer; Radiation
Keywords: DNA; cancer; sequencing technologies; lymphocyte; genomic; loosely ionizing radiation; Linear Energy Transfer; outcome; thoracic radiotherapy
MeSH Terms: conditions — Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Interventional Arm (Experimental)
  Interventions: Radiation: genomic alterations

INTERVENTIONS:
Radiation: genomic alterations — Alteration of the genome under radiotherapy

SUMMARY:
The long-term goal is to define "signatures" in the form of genomic changes through sequence analyses of genomic DNA using modern Next Generation Sequencing (NGS) methods, which

1. determine the radiation exposure of humans.
2. provide information about the exposure (dose).
3. determine the radiation quality.
4. predict the repair capacity and radiation resistance of an individual.

DETAILED DESCRIPTION:
The planned research work will investigate structural changes in DNA caused by loosely ionizing and high-LET (Linear Energy Transfer) radiation as well as their attribution to double-strand break repair pathways, which will be analysed in parallel using modern microscopy methods. Our aim is to incorporate sequencing technologies into the spectrum of methods used in radiation research and radiation protection. It is important for us to consider the practical requirements of radiation protection and to extend our experimental approaches to cell types relevant to radiation protection. For this reason, we have now created a separate work program that will focus specifically on sequence analyses in irradiated human lymphocytes. The aim is to successfully transfer the experimental approaches and bioinformatic analyses established in previous experiments in human skin fibroblasts to lymphocytes. Subjects can donate blood samples on a voluntary basis at predetermined times. Only subjects without previous radiotherapy, chemotherapy, immunotherapy, targeted therapy, etc. and without a previous tumor diagnosis in the medical history and in good performance status (ECOG 0-1) will be included.

ELIGIBILITY:
Inclusion Criteria:

ECOG 0/1 no prior treatment no prior cancer diagnosis thoracic or head and neck cancer

Exclusion Criteria:

prior treatment (chemotherapy, radiotherapy, etc.) prior cancer diagnosis

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2024-06-01 (Actual); Primary Completion 2025-12-15 (Estimated); Study Completion 2030-01-15 (Estimated)

PRIMARY OUTCOMES:
Alteration of the genome under radiotherapy | 5 years
  Radiotherapy of patients, quantitative tissue sampling, cell culture survival rate and mitotic index after predifined radiation treatment, Incidence of the sample and percentage

SECONDARY OUTCOMES:
Overall Survival | 5 years
  Overall Survival
Progression Free Survival | 5 years
  Progression Free Survival
Radiation induced changes in the genome | 2 months to 5 years
  Radiation induced changes in the genome analyzing human skin fibroblasts and lymphocytes:
  translocations that permitted cell division andm mismatch repair of radiation-induced DNA damage (PCR and M-FISH), Incidence of the sample and percentage

CONTACTS AND LOCATIONS:
Locations (1):
- Department for Radiotherapy, University Hospital Essen, National Center for Tumor Diseases (NCT) West, Essen, Germany / NRW, Germany

IPD SHARING:
Plan to Share IPD: No